CLINICAL TRIAL: NCT03162978
Title: Effect of Outcome Expectations on Psychological and Physiological Responses to Interval Exercise Training
Brief Title: Sprint to Fitness: Effect of Outcome Expectations on Responses to Interval Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GFHNRC407
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Overweight; Obesity
Keywords: Exercise; behavior economics
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT + POE (Experimental): High-intensity interval training (HIIT) plus positive outcome expectations (POE) from participating in the exercise program.
  Interventions: Other: HIIT + POE
- HIIT only (Experimental): High-intensity interval training (HIIT) only.
  Interventions: Other: HIIT only

INTERVENTIONS:
Other: HIIT + POE — Subjects will participate in high-intensity interval training (HIIT) with an additional treatment component to increase positive outcome expectations (POE) of exercise.
  Arms: HIIT + POE
Other: HIIT only — Subjects will participate in high-intensity interval training (HIIT) only.
  Arms: HIIT only

SUMMARY:
The purpose of this study is to research the effects of exercising at high intensities for short periods of time on exercise tolerance and motivation.

DETAILED DESCRIPTION:
The proposed research will investigate whether adding a treatment component that focuses on positive outcome expectations of a high-intensity interval training (HIIT) intervention produces greater improvements in psychological and physiological study outcomes. This project will yield empirical evidence that will inform how to help Americans meet physical activity guidelines; how to develop exercise programs that are more likely to promote exercise as a habit; and maintenance of health and a healthy body weight.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index of 25-35 kg/m2
* Sedentary (not regularly engaging in exercise more than once per week)
* Weight stable (have not lost or gained over 10 pounds of body weight in the past 3 months)

Exclusion Criteria:

* Taking any medications that affect energy expenditure or treat high blood pressure
* Tobacco use
* Pregnant or breastfeeding or plan to become pregnant in the next 3 months
* Have any medical conditions that prevent subject from safely exercising (e.g., orthopedic injuries, cardiovascular, liver, endocrine, or pulmonary diseases)
* Resting systolic blood pressure ≥ 140 mmHg
* Resting diastolic blood pressure ≥ 90 mmHg
* Non-fasting plasma glucose of ≥ 200 mg/dl

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Change in relative reinforcing value (RRV) of physical activity | Week 0, Week 6, Week 10
  RRV of physical activity will be assessed by evaluating the number of responses (mouse button presses) a subject is willing to complete to gain access to physical activity or a sedentary alternative.
Changes in preference for intense physical activity and tolerance for exercise discomfort | Week 0, Week 6, Week 10
  Changes in preference for intense physical activity and tolerance for exercise discomfort will be assessed by self-report questionnaire responses to the Preference for and Tolerance of the Intensity of Exercise Questionnaire (PRETIE-Q). The PRETIE-Q measures preference for high intensity vs. low intensity exercise and ability to persist or tolerate the discomfort associationed with intense exercise. The PRETIE-Q consists of two subscales: Preference for Exercise Intensity and Tolerance of Exercise Intensity. Each subscale has 8 items rated on a 5 point response scale (range 8 - 40). Higher scores indicate greater preference for intense exercise and/or greater tolerance for exercise discomfort. Total scale scores are not used. Scale averages will be used.

SECONDARY OUTCOMES:
Change in minutes of physical activity, as assessed by activity tracker | Week 0, Week 6, Week 10
  Minutes of physical activity will be assessed by having participants wear an Actigraph accelerometer for 7 days (minimum 10 hours per day) on the right hip.
Changes in quadriceps and hamstring (thigh muscle) strength assessed separately on each leg | Week 0, Week 6, Week 10
  After range of motion is determined, participants will engage in a series of extensions and flexions in which maximum velocity is set at 60°, 180°, and 300°.s±1 to determine each leg's peak torque as assessed by isokinetic dynamometer testing (Biodex System 4 Pro).
Changes in aerobic fitness, as assessed using the Standardized Exponential Exercise Protocol (STEEP) | Week 0, Week 6, Week 10
  After a brief warm-up, participants will pedal on an ergometer 75-85 revolutions per minute (RPMs) at low resistance of approximately 2 metabolic equivalent of task (METs). The resistance will increase by 15% per minute until respiratory exchange ratio (RER) exceeds 1.0, maximum oxygen consumption (V02 max) is reached, or participant can no longer maintain pedaling speed.
Changes in anaerobic power, as during a Wingate anaerobic power exercise test | Week 0, Week 6, Week 10
  Following a brief warm-up, participants will be instructed to pedal on an ergometer as hard and as fast as they can for 30 seconds at a resistance of 1 watt·kilogram-1, followed by a cool-down period. Changes in anaerobic power, will be as assessed by as changes in power outputs in watts (rpm·braking force).
Changes in fat mass as assessed by dual energy x-ray absorptiometry (DXA) scans | Week 0, Week 6, Week 10
  Participants will be instructed to lie supine with hands by their sides on a GE Lunar iDXA machine for a full-body x-ray scan which will measure grams and percentage changed in fat mass.
Changes in fat-free lean mass as assessed by DXA scans | Week 0, Week 6, Week 10
  Participants will be instructed to lie supine with hands by their sides on a GE Lunar iDXA machine for a full-body x-ray scan which will measure grams and percentage changed in fat-free lean mass.
Changes in tolerance for physical pain and discomfort | Week 0, Week 6, Week 10
  Changes in preference for tolerance for physical pain and discomfort will be assessed by self-report questionnaire responses to the Discomfort Intolerance Scale (DIS). This scale measures individual differences in ability to tolerate uncomfortable sensations. There are 7 items total. Although there are two subscales (measure ability to tolerate discomfort / pain and avoidance of physical discomfort) only total scores will be used. There are 7 items total. Items are scored 0 - 6 (total range 0 - 42), with higher scores indicating greater ability to tolerate physical discomfort. Average score on the total scale will be used.
Changes in perceived support for physical activity from friends and family members | Week 0, Week 6, Week 10
  Changes perceived support for physical activity from friends and family members will be assessed by self-report questionnaire responses to the Social Support and Exercise Survey. This questionnaire measures 13 items are scored on a scale of 1 - 5, with higher scores indicating greater perceived support. Total scores will be used, with ranges from 13 - 65. Higher scores indicate greater perceived support. Average score for the total scale will be used. Items may be answered twice, once for family members and once for friends.
Changes in perceptions of how much exercise satisfies autonomy, relatedness, and competence needs | Week 0, Week 6, Week 10
  Changes in perceptions of how much exercise satisfies autonomy, relatedness, and competence needs will be assessed by self-report questionnaire responses to the Psychological Need Satisfaction in Exercise Scale. This scale measures how much the psychological needs of autonomy, relatedness, and competence are satisfied during exercise. There are three subscales: autonomy, relatedness, and competence. Each subscale has 6 items rated on a 6-point scale. Higher scores indicate greater amounts of the construct. Total subscale scores may range from 6 to 36. Subscale averages will be used in analyses.
Changes in intrinsic, external, interrogated, identified, introjected and amotivation for physical activity | Week 0, Week 6, Week 10
  Changes in intrinsic, external, interrogated, identified, introjected and amotivation for physical activity will be assessed by self-report questionnaire responses to the Behavioral Regulation in Exercise, 3rd Edition (BREQ-3).This scale measures how much exercise behavior is driven by intrinsic motivation, external motivation, interrogated motivation, identified motivation, introjected motivation, and amotivation (lack of motivation). There are 6 subscales with 4 items each: intrinsic, external, interrogated, identified, introjected, and amotivation. Items are measured on a 5-point scale, where higher scores indicated greater amounts of the construct. Subscale scores may range from 4 to 20. Average subscale scores will be used in analyses.
Changes in how enjoyable physical activity is perceived to be | Week 0, Week 6, Week 10
  Changes in how enjoyable physical activity is perceived to be will be assessed by self-report questionnaire responses to the Physical Activity Enjoyment scale (PACES). This scale measures how enjoyable or unenjoyable physical activity is perceived to be. The measure consists of 18 questions and no subscales. Each question is measured on a 7-point scale, where higher scores indicate greater enjoyment. Total scores may range from 18 to 126. Average score will be used.
Changes in perceived effort expended during exercise | Week 0, Week 6, Week 10
  Changes in perceived effort expended during exercise will be assessed by self-report questionnaire responses to the Borg Rating of Perceived Exertion Scale. This scale measures perceived physical exertion during exercise. There is only 1 item and no subscales. Scores may range from 0 to 10, with higher scores indicating greater perceived exertion. The total score will be used in analyses.
Changes in perceived pain/discomfort during exercise | Week 0, Week 6, Week 10
  Changes in perceived pain/discomfort during exercise will be assessed by self-report questionnaire responses to the Numeric Ratings Pain Scale. This single item scale measures muscle pain/discomfort associated with physical activity. There are no subscales. Scores may range from 0 to 11, with higher scores indicating greater pain/discomfort. The total score will be used in analyses.
Changes in perceived ability to continue exercise long-term | Week 0, Week 6, Week 10
  Changes in perceived ability to continue exercise long-term will be assessed by self-report questionnaire responses to the Barriers Self-Efficacy Scale (BARSE). This scale measures perceived ability to continue meeting exercise guidelines over the next 1 to 8 weeks. There are no subscales. 8 items are measured on an 11-point scale where higher scores indicate greater certainty in ability to complete exercise. Average score will be used in analyses.
Changes in perceived ability to stick to an exercise routine | Week 0, Week 6, Week 10
  Changes in perceived ability to stick to an exercise routine will be assessed by self-report questionnaire responses to the Exercise Confidence Survey. This scale measures perceived confidence in ability to make time for exercise and persist in an exercise routine. There are 2 subscales: sticking to it (8 items) and making time for exercise (4 items). Items are measured on a 5-point scale where higher scores indicate greater confidence. Total scores may range from 8-40 (sticking to it) or 4-20 (making time). Average subscale scores will be used in analyses.

CONTACTS AND LOCATIONS:
Overall Officials: James N Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/

DOCUMENTS (1):
  • Informed Consent Form (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT03162978/ICF_000.pdf